CLINICAL TRIAL: NCT05411952
Title: The Effect of Family-Based Behavioral Medical Nutrition Therapy Education on Nutritional Status and Metabolic Control in Children and Adolescents With Type 1 Diabetes
Brief Title: Family-Based Behavioral Medical Nutrition Therapy Education in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hasan-Kalyoncu-UnivHulyaYilmaz
Record Dates: First submitted 2022-05-30; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Type1diabetes
Keywords: Type 1 diabetes, nutrition education, metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: The sample of the study was consisted of 75 (male= 36, female= 39) children and adolescents in total, including Intervention 1 group (n=25), Intervention 2 (n=25) group and Control (n=25) group determined by double-blind, stratified, random method.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- education-mother and child dyad (Experimental): Mother and child dyad have received dietary intervention for 6 months
  Interventions: Other: Medical nutrition therapy and carbohydrate counting education
- education-only child (Experimental): Children have received dietary intervention for 6 months. But their mothers didn't receive any dietary intervention
  Interventions: Other: Medical nutrition therapy and carbohydrate counting education
- control (Experimental): Control group did't receive any dietary intervention during the study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Medical nutrition therapy and carbohydrate counting education — Children and their mothers have received family-based behavioral medical nutrition therapy and carbohydrate counting education for 6 months by trained dietitian
  Arms: education-mother and child dyad
Other: Medical nutrition therapy and carbohydrate counting education — Only children have received family-based behavioral medical nutrition therapy and carbohydrate counting education for 6 months by trained dietitian
  Arms: education-only child
Other: No intervention — Control group didn't receive any intervention by trained dietitian. Furthermore they continued their routine health controls.
  Arms: control

SUMMARY:
Type 1 Diabetes Mellitus (T1DM) is a heterogeneous condition and is an absolute insulin deficiency resulting from autoimmune-mediated destruction of pancreatic β-cells (1). The incidence of T1DM has been increasing globally since the 1950s, particularly in children, with an average annual increase of 3-4% over the past three decades.Despite the advances in medical treatment and technology, nutritional therapy continues to be the main component of diabetes treatment. Medical nutrition further improves metabolic control outcomes when T1DM care is combined with other treatments.This study was conducted to examine the effect of family-based behavioral medical nutrition therapy training on nutritional status and metabolic control in children and adolescents with Type 1 diabetes.

DETAILED DESCRIPTION:
The research was carried out with children and adolescents aged 8-18 years who were followed up with the diagnosis of Type 1 Diabetes Mellitus in Gaziantep Cengiz Gökçek Gynecology and Pediatrics Hospital. The sample of the study was consisted of 75 (male= 36, female= 39) children and adolescents in total, including Intervention 1 group (n=25), Intervention 2 (n=25) group and Control (n=25) group determined by double-blind, stratified, random method. Medical nutrition therapy and carbohydrate counting training were given to mothers and children in the Intervention 1 group, and only to children and adolescents in the Intervention 2 group. The control group did not receive medical nutrition therapy and carbohydrate counting training. At the beginning (0. month) and at the end (6. month) of the study, 3 consecutive day/24-hour food consumption records and anthropometric measurements of the individuals were assessed, BMI z-scores and height z-scores were calculated, Mediterranean Diet Quality Index Scale (KIDMED), Diabetes Eating Problems Survey-Revised (DEPS-R), Physical Activity Questionnaire for Children and Adolescents (PAQ-C and PAQ-A) were administered and Healthy Eating Index 2015 (HEI-2015) scores were calculated. Routinely assessed blood findings of the individuals were checked at the beginning (0. month), 3rd month and 6th month of the study.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years old,
* Being diagnosed with T1DM for at least ≥1 year, maximum ≤5 years,
* Latest HbA1c ≥6.5% - <13.5%,
* Receiving intensive insulin therapy (at least 3 times a day bolus and 1 time basal insulin administration or using an insulin pump),
* No communication problems
* Children and adolescents without any other disease accompanying diabetes were included in the study.

Exclusion Criteria:

* Celiac, cystic fibrosis etc. with gastrointestinal diseases,
* Using any drug that may affect glucose metabolism,
* Switched from an insulin pen to an insulin pump in less than 6 months,
* Involved in any other intervention work in the last 6 months,
* and individuals with communication problems were not included in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change in mean of HbA1c from baseline to 6 months | 6 months
  All data were analysed by using IBM SPSS Statistics 26 and significance was defined as p< 0.05

SECONDARY OUTCOMES:
Change in mean of Healthy Eating Index 2015 (HEI-2015) score from baseline to 6 Months | 6 months
  All data were analysed by using IBM SPSS Statistics 26 and significance was defined as p< 0.05
Change in mean of Mediterranean Diet Quality Index Scale (KIDMED) from baseline to 6 Months | 6 months
  All data were analysed by using IBM SPSS Statistics 26 and significance was defined as p< 0.05

CONTACTS AND LOCATIONS:
Overall Officials: Gulden KOKSAL, Prof., Study Director — Hasan Kalyoncu University
Locations (1):
- Gaziantep Cengiz Gokcek Gynecology and Pediatrics Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No